CLINICAL TRIAL: NCT06581523
Title: A Feasibility and Efficacy Study of a Breathwork and Meditation Intervention (SKY Breath) on the Psychophysiological Well-Being of Individuals With Parkinson's Disease (iPD) and Their Care Partners
Brief Title: Efficacy of a Breathwork Practice (SKY) on Well-Being of Individuals With Parkinson's Disease (iPD) and Care Partners
Acronym: SKYforiPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-434-NSU
Record Dates: First submitted 2024-08-29; First posted 2024-09-03 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Sudarshan Kriya Yoga; SKY Breath and Meditation; Care Partner of Individuals with Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: The SKY Breath and Meditation intervention will be for both the individuals with Parkinson's Disease and their care partners.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual with Parkinson's Disease (Experimental): The intervention is the Sudarshan Kriya Yoga or SKY Breath and Meditation Practice. This will be taught over a 10-12 hour period, 2.25 hours for 4 early mornings. The participants will practice 6 days a week (a 35-45 minute practice)for a total of 8 weeks.
  Interventions: Behavioral: SKY Breath and Meditation
- Care Partner of Individual with Parkinson's Disease (Experimental): The intervention is the Sudarshan Kriya Yoga or SKY Breath and Meditation Practice. This will be taught over a 10-12 hour period, 2.25 hours for 4 early mornings. The participants will practice 6 days a week (a 35-45 minute practice)for a total of 8 weeks.
  Interventions: Behavioral: SKY Breath and Meditation

INTERVENTIONS:
Behavioral: SKY Breath and Meditation — SKY Breath and Meditation is a unique breath-based technique that uses cyclical, rhythmic patterns of breath to bring the mind and body effortlessly into meditation. It has been empirically validated and holds distinct advantages over other forms of meditation.
  Other Names: Sudarshan Kriya Yoga; SKY Breath

SUMMARY:
The goal of this feasibility study and clinical trial is to learn if an evidenced-based breathwork and meditation intervention (SKY Breath) will improve the mental and physical well-being of individuals with Parkinson's Disease (iPD) in stages 1, 2, and 3, under the age of 75 and their care partners. The main questions it aims to answer are:

* Objective 1: Can the SKY Breath practice be designed and implemented to specifically cater to the unique needs of individuals with Parkinson's Disease and their care partners.
* Objective 2: Will the SKY Breath practice decrease stress levels (a contributor to increasing PD symptoms) for individuals with Parkinson&amp;#39;s Disease (iPD) and their care partners as measured through self-reported surveys to improve overall well-being and quality of life.
* Objective 3: Will the SKY Breath practice in part alleviate the emotional stress and physical burden experienced by care partners of PD patients, promoting their resilience and well-being.

Participants will be asked to learn the SKY Breath and Meditation practice over the course of 4 days (2.25 hours each morning), practice SKY every day for 4 weeks and keep a log of time spent doing SKY. The participants will complete a series of surveys before learning the practice and then after at weeks 1, 4 and 8. The series of surveys will take about 20 minutes.

DETAILED DESCRIPTION:
Protocol Summary

Introduction: Parkinson's Disease (PD) is a neuro-degenerative disease and movement disorder with no known cure. Symptoms include tremor and neuro-psychiatric issues. Stress significantly exacerbates symptoms of PD. This study aims to determine the feasibility and efficacy of an evidence-based stress reduction and resilience building breathwork intervention named Sudarshan Kriya Yoga (SKY) Breath and Meditation (SKY Breath) to improve the psycho-physiological wellbeing in a cohort of community dwelling individuals diagnosed with Parkinson's Disease (iPD).

Methodology: This mixed methodology feasibility study will evaluate the tremor, gait, mental wellbeing of a cohort of patients from several organizations with iPD. Measures of motor and non-motor symptoms will be tested before and after the intervention. The standardized program will be modified according to the level of iPD disability and limitation. Data is stratified according to disability level. 20 iPD and 20 care partners will be consented for participation.

Active Learning Phase 1: A 10-12 hour active learning phase (4 day morning program) will be presented. The length of this phase will be determined upon iPD participant stamina. Participants will be given a home practice to complete with an audiotape and a handout as a supplement. When necessary, the SKY Breath practice can be broken up to accommodate a schedule. This will encourage as many individuals as possible to participate. A parallel course will be given to the care partners.

Phase 2:This includes daily personal home practice taking about 25 minutes, which can be done independently or online with instructor. There is also once weekly instructor guided session online lasting approximately 45 minutes. And one weekly session in-person, lasting 75 minutes. IPD Measures standardized measures of PD symptoms motor and non-motor symptoms and Quality of Life (QoL) care partners receive QoL, stress and resilience measured. Participants will be evaluated pre-intervention, post week 2 and 8.

Recruiting will be done at a Gym teaching Rock Steady Boxing/Coral Springs, Cleveland Clinic and at the David Posnack JCC as well as through the NSU Clinics (Flyers will be placed so that existing patients from the Department of Physical Therapy at NSU can inquire and be recruited). Results: Data will be analyzed using repeated measure ANOVA, with post hoc analysis of interactions between outcomes. Qualitative data will be scored for themes.

3. Background / Aims

1. Purpose Statement: This study aims to determine the feasibility and efficacy of an evidence-based stress reduction/resilience building breathwork intervention named Sudarshan Kriya Yoga Breath and Meditation (SKY Breath) to improve the psycho-physiological wellbeing in a cohort of community dwelling individuals diagnosed with PD (iPD) and their care partners.
2. Objectives +/- Hypotheses:

Objective 1: Alleviate Stress for Parkinson's Disease (PD) Patients and Care partners Implement a SKY breath intervention to actively minimize stress levels in both PD patients and their care partners, contributing to an improved overall well-being and quality of life.

Objective 2: Develop Targeted Programs for PD Patients Design and implement effective and tailored programs specifically catering to the unique needs of PD patients and their care partners. Ensuring a comprehensive, cost effective, self-empowering treatment protocol that will contribute to improving the overall well-being and quality of life of the patients.

Objective 3: Relieve Burden on Care partners Introduce interventions and support mechanisms to alleviate the emotional and physical burden experienced by care partners of PD patients, promoting their resilience and well-being.

Objective 4: Alleviate Strain on the Healthcare System Implement strategies that reduce the strain on the healthcare system by enhancing the self-management capabilities of PD patients and their care partners, leading to potentially fewer hospital visits and resource utilization.

Objective 5: Establish a Compassionate and Comprehensive Model for PD Care Develop and propose a model for PD care that prioritizes compassion and comprehensiveness, serving as a potential blueprint for future healthcare practices in Parkinson's Disease adjunctive management.

Study Design (including Basic Timeline)

1. Methodology This mixed methodology feasibility study will evaluate the tremor, balance mental wellbeing of a cohort of patients from several organizations that have a group of PD patients. The study will consent and enrolls 20 iPD and 20 care partners. The iPD will have their disease stage evaluated using the Hoehn and Yahr scale.

   Both the iPD and their care partners will be evaluated pre and post intervention on measures of anxiety and depression to include the Perceived Stress Scale (PSS). Measures of psycho-social wellbeing will also be measured. The research will also evaluate specific measures of function of for the iPD using the The International Parkinson and Movement Disorder Society sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS). All aspects of the SKY standardized program will be modified according to the level of disability and limitation. The other measures that will be used are:
   * Positive and Negative Affect Scale (PANAS)
   * Parkinson's Anxiety Scale
   * Parkinson's Disease Care Giver Burden Questionnaire (PDCG)
   * Parkinson's Fatigue Scale
   * Parkinson's Disease Quality of Life (PDQ-39)

   The data will be stratified according to their level of disability and physical limitation.

   After the pre-testing evaluation is done prior to the SKY Breath Intervention being taught to the iPD and their care partners at one of potentially three sites (RAW Kickboxing GYM, David Posnack Jewish Community Center, DPJCC), Cleveland Clinic).

   There are two phases to the SKY Breath intervention include 1). Phase 1: The Active Learning Phase and 2). Phase 2: The Booster and reinforcement sessions.

   Active Learning Phase:

   A 10-12 hour active learning phase (4 day morning program 2.25 hours each day) will be presented. The length of the active learning phase that is presented will be determined depending on the stamina of the participants. The PD patients will be given a home practice to complete with an audiotape. A handout will be given to the participants as a supplement. When necessary, the SKY Breath practice can be broken up to accommodate a schedule. This will encourage as many individuals as possible to participate.

   A parallel course will be given to the Care partners.

   Phase 2:

   This includes daily personal home practice and twice weekly instructor guided group sessions. One weekly session will be online, lasting approximately 45 minutes. The second weekly session will be in-person, lasting approximately 75 minutes.

   The validated measures will be the standardized measures of PD symptoms The International Parkinson and Movement Disorder Society sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) capturing the disease stage with the modified Hoehn and Yahr Scale that is part of the MDS-UPDRS. This is in addition to the:
   * Positive and Negative Affect Scale (PANAS)
   * Parkinson's Disease Anxiety Scale
   * Parkinson's Fatigue Scale
   * Parkinson's Disease Quality of Life Scale (PDQ-39)
   * Perceived Stress Scale (PSS)

   Care partners will be evaluated with:
   * Positive and Negative Affect Scale (PANAS)
   * Parkinson's Disease Care Giver Burden Questionnaire (PDCG)
   * Perceived Stress Scale (PSS)

   The PD individuals will be evaluated prior to learning the SKY Breath Practice and then 1 week, 4 weeks and 8 weeks post-intervention. The participants will need to practice 6 days a week that will be lead by a qualified instructor. The practice will be lead once a week on-line and once a week in person. (One practice will be done in the early morning by Zoom and one will be done on a weekend day in the afternoon).
2. Schedule of Events Weeks 1 - 2: Collaborative development of recruiting materials and preparation of Institutional Review Board (IRB) application.

Week 3: Submission of IRB application, recruiting of Nova Southeastern University (NSU) students as Research Assistants and assistant coordinators

Weeks 4-6: Training of NSU students for screening and administration of the test instruments.

Weeks 6- 11: Active recruiting, screening, and consenting of iPD and their care partners(assuming IRB approval)

Weeks 10 - 11: baseline data collection (while to be conducted online)

Week 11: Phase 1 of SKY breath meditation intervention (3 to 4 of 2 ½- 3 hours each sessions on consecutive mornings in person)

Week 12 - 19: Once weekly in person group SKY booster session lasting 75 to 90 minutes, plus one online group SKY practice lasting 60 minutes.

Week 14:1st posttest

Week 20: Final posttest

Week 21: Focus group for iPD group and separate focus group for care partners

Weeks 22- 23 Data analysis

ELIGIBILITY:
Inclusion Criteria:

Individuals with Parkinson's Disease (iPD) Inclusion Criteria: An individual with a formal diagnosis of iPD that:

* are in stages 1, 2, or 3
* are at least 18 years of age
* are no older than 75 years of age
* can understand, read, write and speak English at a 5th grade level
* that have access to zoom sessions online via laptop, ipad or other mobile device
* are able to secure reliable transportation for themselves.

Care Partner of the individuals with Parkinson's Disease (iPD) Inclusion Criteria: Individuals who:

* are a care partner for an individual with Parkinson's Disease but are not paid professional givers of care
* are at least 18 years of age or older
* are able to secure reliable transportation for themselves and for the Individual with Parkinson's Disease
* can understand, read, write and speak English at a 5th grade level
* has access to zoom sessions online via laptop, iPad or other mobile device.

Exclusion Criteria:

Individuals with Parkinson's Disease (iPD): An individual who

* has been diagnosed with Parkinson's Disease that is in stages 4 or 5 of the disease
* is younger that age 18 or older than age 75
* has bipolar disorder
* has seizure disorder
* has schizophrenia or schizoaffective disorder
* has active substance use
* has uncontrolled hypertension
* has cognitive impairment that prevents them from memorizing (remembering) the steps to complete the daily breath and meditation practice or completing the survey instruments, or has difficulty following sequential directions of the breathing practice
* cannot understand, read, write and speak English at a 5th grade level
* does not have access to zoom sessions online via laptop, iPad or other mobile device
* can not secure transportation to the site for the training of the breath and meditation practice

Care partner of the Individuals with Parkinson's Disease (iPD): Individuals who:

* are paid professional givers of care
* are under the age of 18
* an emancipated minor
* have bipolar disorder
* have seizure disorder
* have schizophrenia or schizoaffective disorder
* have active substance use
* have uncontrolled hypertension
* are not able to secure reliable transportation for themselves
* cannot understand, read, write and speak English at a 5th grade level
* does not have access to access to zoom sessions online via laptop, iPad or other mobile device.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-19 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Stress management for Individuals with Parkinson's Disease | Pre-intervention, and 2 weeks, 4 weeks, 8 weeks post intervention
  Improving the feelings of pressure and overwhelm measured before and after intervention from self-reported stress scales. Individuals with Parkinson's Disease evaluated on:
  * Parkinson's Disease Anxiety Scale- Scoring 0-48. Higher score=greater anxiety.
  * Perceived Stress Scale (PSS) -Scores from 0-40; higher scores=higher perceived stress.
Stress management for Care Partners of Individuals with Parkinson's Disease | Pre-intervention, and 2 weeks, 4 weeks, 8 weeks post intervention
  Improving the feelings of pressure and overwhelm measured before and after intervention from self-reported stress scales. Care partners evaluated on:
  * Parkinson's Disease Care Giver Burden Questionnaire (PDCG) -Scoring 0-20=little/no burden;21-40=mild/moderate burden;41-60=moderate/severe burden;61-88=severe burden.
  * Perceived Stress Scale (PSS) -Scoring 0-40; higher scores=higher perceived stress.
Psycho-social well-being management for Individuals with Parkinson's Disease | Pre-intervention, and 2 weeks, 4 weeks, 8 weeks post intervention
  Improving the general perceived mental health and well-being of individuals measured from self-reported scales. Individuals with Parkinson's Disease evaluated on:
  * Positive and Negative Affect Scale (PANAS)- Scoring 10-50 both sets. Total positive score, higher score=more positive affect. Total negative score, a lower score= less negative affect.
  * Parkinson's Fatigue Scale-Scoring 0-36. Total score of less than 36=may not be suffering from fatigue.
  * Parkinson's Disease Quality of Life Scale (PDQ-39)-Scoring 0-260; 0=no disability; 260=total disability.
Psycho-social well-being management for Care Partners of Individuals with Parkinson's Disease | Pre-intervention, and 2 weeks, 4 weeks, 8 weeks post intervention
  Improving the general perceived mental health and well-being of individuals measured from self-reported scales. Care partners evaluated on:
  * Positive and Negative Affect Scale (PANAS)- Scoring 10-50 for both sets. Total positive score, a higher score=more positive affect. Total negative score, a lower score= less negative affect.
  * Parkinson's Disease Care Giver Burden Questionnaire (PDCG) -Scoring 0-20=little/no burden;21-40=mild/moderate burden;41-60=moderate/severe burden;61-88=severe burden.
Parkinson's Disease Symptom management/Relief | Pre-intervention, and at 2 weeks, 4 weeks and 8 weeks post intervention
  Improving the symptoms of gait, balance, energy levels in individuals with Parkinson's Disease as measured from
  * the Hoehne and Yahr Scale taken as part of The International Parkinson and Movement Disorder Society sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS).
  * Score range: 0-52, 10 and below is mild, 22 and above is severe. Part II: Motor experiences of daily living: 13 items. Score range: 0-52, 12 and below is mild, 30 and above is severe.

CONTACTS AND LOCATIONS:
Overall Officials: Venetia Bennett, BS, MS, PhD, Principal Investigator — Nova Southeastern University, Kiran Patel College of Osteopathic Medicine
Locations (3):
- United States (3):
  - Raw Kickboxing and Fitness, Coral Springs, Florida
  - David Posnack Jewish Community Center, Davie, Florida
  - Nova Southeastern University, Fort Lauderdale, Florida

IPD SHARING:
Plan to Share IPD: No
There is no plan to share at this point.

REFERENCES:
- [Result] Seppala EM, Bradley C, Moeller J, Harouni L, Nandamudi D, Brackett MA. Promoting Mental Health and Psychological Thriving in University Students: A Randomized Controlled Trial of Three Well-Being Interventions. Front Psychiatry. 2020 Jul 15;11:590. doi: 10.3389/fpsyt.2020.00590. eCollection 2020. PMID 32760296
- [Result] Bayley PJ, Schulz-Heik RJ, Tang JS, Mathersul DC, Avery T, Wong M, Zeitzer JM, Rosen CS, Burn AS, Hernandez B, Lazzeroni LC, Seppala EM. Randomised clinical non-inferiority trial of breathing-based meditation and cognitive processing therapy for symptoms of post-traumatic stress disorder in military veterans. BMJ Open. 2022 Aug 25;12(8):e056609. doi: 10.1136/bmjopen-2021-056609. PMID 36008059
- [Result] Seppala EM, Nitschke JB, Tudorascu DL, Hayes A, Goldstein MR, Nguyen DT, Perlman D, Davidson RJ. Breathing-based meditation decreases posttraumatic stress disorder symptoms in U.S. military veterans: a randomized controlled longitudinal study. J Trauma Stress. 2014 Aug;27(4):397-405. doi: 10.1002/jts.21936. PMID 25158633
- [Result] Korkmaz A, Bernhardsen GP, Cirit B, Koprucu Suzer G, Kayan H, Bicmen H, Tahra M, Suner A, Lehto SM, Sag D, Saatcioglu F. Sudarshan Kriya Yoga Breathing and a Meditation Program for Burnout Among Physicians: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2353978. doi: 10.1001/jamanetworkopen.2023.53978. PMID 38294813
- [Result] Brown RP, Gerbarg PL. Sudarshan Kriya yogic breathing in the treatment of stress, anxiety, and depression: part I-neurophysiologic model. J Altern Complement Med. 2005 Feb;11(1):189-201. doi: 10.1089/acm.2005.11.189. PMID 15750381
- [Result] van Wamelen DJ, Wan YM, Ray Chaudhuri K, Jenner P. Stress and cortisol in Parkinson's disease. Int Rev Neurobiol. 2020;152:131-156. doi: 10.1016/bs.irn.2020.01.005. Epub 2020 Feb 19. PMID 32450994